CLINICAL TRIAL: NCT01036958
Title: Development and Validation of a Symptom Scale for Children With Chronic Graft-Versus-Host Disease
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100019; 10-C-0019
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-02-06

CONDITIONS: Chronic Graft-Versus-Host-Disease
Keywords: Pediatric cGVHD; Response Criteria; Symptoms; Quality of Life; Graft-Versus-Host Disease; GVHD; Pediatric GVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Background:

* Chronic graft-vs-host disease (GVHD) is an important cause of morbidity and mortality in patients undergoing allogeneic bone marrow transplantation. The symptoms of chronic GVHD are similar to those of other autoimmune diseases, and treatment for the pain often involves steroid use that can cause severe side effects over the long term.
* At present, there is no research instrument that measures symptoms in children with chronic GVHD. Treatment practitioners may use one of several pediatric quality of life questionnaires, but because none of these is specific for chronic GVHD each instrument has potential gaps in its ability to assess the full spectrum of problems experienced by children with chronic GVHD. Researchers are interested in developing a better understanding of the disease burden experienced by children and adolescents with chronic GVHD.

Objectives:

- To develop a Pediatric Chronic GVHD Symptom Scale (PCSS) that reliably measures the disease-specific burden of chronic GVHD in children.

Eligibility:

- Children and adolescents 5 to 18 years of age who have undergone prior allogeneic stem cell transplant and have been diagnosed with chronic GVHD that requires treatment.

Design:

* There are two phases to the study; participants will enroll in phase I (question generation) at this time.
* Researchers will interview participants and ask open-ended questions (requiring more than a one- or two-word response) about symptoms that adults with chronic GVHD have found problematic.
* Both parents and children will participate in the interviews, which will be audio-recorded. Depending on the child or adolescent s age, the interviews may be conducted together with the parents or separately.
* No treatment will be given as part of this study.

DETAILED DESCRIPTION:
Background:

* Currently, a large number of children with chronic GVHD have to deal with many years of a disfiguring and painful chronic illness with the side effects of long term steroid use.
* The broad categories of limited and extensive chronic GVHD are recognized by clinicians, but are not particularly useful in clinical practice. Chronic GVHD may involve almost every organ although it most commonly affects skin, eyes, mouth, liver, intestines, lung and musculoskeletal system.
* Recently, there has been a large effort through the NIH Consensus for chronic GVHD to standardize response criteria for patients with chronic GVHD, on clinical trials. Because of the absence of evidence suggesting which response criteria truly correlates with improvement, the NIH Consensus Panel has recommended following not only physical signs of chronic GVHD, but also symptoms of GVHD.

Primary Objective:

- Develop a Pediatric Chronic GVHD Symptom Scale (PCSS) that reliably measures the disease specific burden of chronic GVHD in children.

Secondary Objectives:

* Correlate high and low scores on the PCSS with standard quality of life measures.
* Determine using the Rasch measurement model whether the PCSS has sufficient sensitivity to change for the scale to be useful in clinical intervention trials.

Eligibility:

* Children of 5 to 18 years of age, who have undergone prior allogeneic stem cell transplant
* Clinical diagnosis of chronic GVHD with need for systemic treatment
* No evidence of primary disease relapse
* Must be willing to sign informed consent, or if applicable, child assent

Design:

* With the final goal of developing a scale that is similar in design to the Lee Scale but which measures the symptom burden more specifically for children with chronic GVHD, the study will be conducted in two phases: item generation and psychometric validation.
* In phase I, the local team at each institution will interview participants using a script to identify symptom concerns for pediatric chronic GVHD patients. Based on interviews, we will decide whether to test different scales for the different age groups, or a single scale for all.
* Data from Phase II will be used to finalize and validate the pediatric symptom scale, through the assessment of test-retest characteristics, use of item reduction, examination of construct validity, internal consistency, convergent and divergent validity, and evaluation of sensitivity to change.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Children of 5 to 18 years of age, who have undergone prior allogeneic stem cell transplant.
* Clinical diagnosis of chronic GVHD with need for systemic treatment.
* No evidence of primary disease relapse.
* Must be willing to sign informed consent, or if applicable, child assent.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2009-11-25; Study Completion 2018-02-06

PRIMARY OUTCOMES:
Develop pediatric cGVHD symptom scale | 24 months

SECONDARY OUTCOMES:
Rasch measurement model, determine sensitivity to use in clinicalintervention trials | 24 months
Correlate scores with QOL measures | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori Wiener, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Champlin RE, Gale RP. The early complications of bone marrow transplantation. Semin Hematol. 1984 Apr;21(2):101-8. No abstract available. PMID 6377500
- [Background] Thomas E, Storb R, Clift RA, Fefer A, Johnson FL, Neiman PE, Lerner KG, Glucksberg H, Buckner CD. Bone-marrow transplantation (first of two parts). N Engl J Med. 1975 Apr 17;292(16):832-43. doi: 10.1056/NEJM197504172921605. No abstract available. PMID 234595
- [Background] Sullivan KM, Parkman R. The pathophysiology and treatment of graft-versus-host disease. Clin Haematol. 1983 Oct;12(3):775-89. doi: 10.1016/s0308-2261(83)80010-1. PMID 6315285